CLINICAL TRIAL: NCT02244619
Title: Randomized, Double-Blind, Study Comparing Oral Acetaminophen Plus Intravenous (IV) Placebo to Oral Placebo Plus IV Acetaminophen Given Perioperatively for Controlling Pain in the 24hr Post-op Period After Total Hip or Knee Joint Replacement
Brief Title: PO vs. IV Acetaminophen Given Perioperatively for 24 hr Post-op Pain Control Following Total Hip or Knee Replacement
Acronym: KHEA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kettering Health Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: KMCPH-13-001
Record Dates: First submitted 2014-09-16; First posted 2014-09-19 (Estimated); Results first posted 2017-07-24 (Actual); Last update posted 2017-07-24 (Actual); Status verified 2017-07

CONDITIONS: Post-op Pain
Keywords: Hip replacement; Knee replacement; randomized trial; acetaminophen; post-op pain management
MeSH Terms: conditions — Pain, Postoperative | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral acetaminophen (Active Comparator): Subjects receive 2 capsules each containing Tylenol 500 mg caplets. The test article administration will be initiated 60 minutes (± 15 minutes) prior to the scheduled surgery start time.
  Interventions: Drug: Oral acetaminophen
- IV acetaminophen (Active Comparator): Subjects receive Ofirmev 1000 mg in 100 ml Normal Saline IV infusion. The test article will be given perioperatively at the discretion of the attending anesthesiologist.
  Interventions: Drug: IV acetaminophen

INTERVENTIONS:
Drug: Oral acetaminophen — Subjects randomized to the Oral acetaminophen arm will receive 2 Tylenol 500mg capsules. In this study, one arm receives an oral form of active medication and one arm receives an IV form of active medication. To keep the subject and study personnel blinded, subjects receiving Oral acetaminophen will also receive 100ml of IV Normal Saline similar to the delivery method of the IV acetaminophen arm. The Normal Saline IV placebo will be given not as an intervention but rather as a method to maintain study integrity.
  Other Names: Tylenol
  Arms: Oral acetaminophen
Drug: IV acetaminophen — Subjects randomized to the IV acetaminophen arm will receive Ofirmev 1000mg in 100ml Normal Saline IV plus 2 placebo capsules. In this study, one arm receives an oral form of active medication and one arm receives an IV form of active medication. To keep the subject and study personnel blinded, subjects receiving IV acetaminophen will also receive 2 placebo capsules similar to the delivery method of the oral acetaminophen arm. The placebo capsules will be given not as an intervention but rather as a method to maintain study integrity.
  Other Names: Ofirmev
  Arms: IV acetaminophen

SUMMARY:
The purpose of the study is to evaluate post-op pain requirements in patients undergoing hip or knee replacement surgery who perioperatively receive either Oral acetaminophen or IV acetaminophen

DETAILED DESCRIPTION:
Subjects will be randomized to receive perioperative dosing of either:

1. Oral acetaminophen (Tylenol) 1000mg with IV Placebo (100ml Normal Saline), OR,
2. IV acetaminophen (Ofirmev) 1000mg/100ml with Oral Placebo (oral capsules).

Subject pain levels and post-operative opioid use will be tracked for up to 24 hours after surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Able to provide written consent
* Able to read and write in English
* Weighing over 50 kg
* Will undergo total hip or total knee joint replacement

Exclusion Criteria:

* Non-verbal patients
* Unable to use numeric pain scale
* Allergic to the test article
* Documented hepatic impairment or failure
* Current illicit drug use
* Requires traumatic or emergent surgery
* Pregnant women
* Women who are breastfeeding
* Prisoners
* Cognitively impaired requiring Legally Authorized Representative (LAR) or Power of Attorney (POA)
* Unable to swallow oral capsules

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 515 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sidney (Skip) Hickman, RPh, Principal Investigator — Kettering Health Network
Locations (1):
- Kettering Medical Center, Kettering, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oral Acetaminophen | IV Acetaminophen
Started | 249 | 266
Completed | 241 | 245
Not Completed | 8 | 21
Not completed — Did not receive study intervention | 8 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Acetaminophen | IV Acetaminophen | Total
Number analyzed (Participants) | 241 | 245 | 486
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 67.0 [59.5 to 73.0] | 67.0 [60.0 to 72.5] | 67.0 [60.0 to 73.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 148 | 140 | 288
  Male | 93 | 105 | 198
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 7
  Not Hispanic or Latino | 237 | 240 | 477
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 11 | 14
  White | 234 | 230 | 464
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 2 | 0 | 2
Taking medications for chronic pain [Count of Participants; unit: Participants] | 214 | 212 | 426
Oxford score (hip or knee as appropriate) [Mean (Standard Deviation); unit: units on a scale] — 12-item ordinal scales. Each item ranges from 0 (high impairment) to 4 (no impairment). Total score ranges from 0-48 with following interpretation:
  0-19: May indicate severe arthritis.
  20-29: May indicate moderate to severe arthritis.
  30-39: May indicate mild to moderate arthritis.
  40-48: May indicate satisfactory joint function.
  units on a scale | 20.76 (7.5) | 20.19 (7.8) | 20.47 (7.6)
Body mass index [Median (Inter-Quartile Range); unit: lb/in^2x703] — In the study data, BMI ranged from 19 (minimum) to 56 (maximum).
  lb/in^2x703 | 31.9 [28.3 to 37.08] | 32.3 [28.5 to 36.71] | 32.1 [28.4 to 36.8]
Diabetes [Count of Participants; unit: Participants] | 48 | 50 | 98
Stroke [Count of Participants; unit: Participants] | 5 | 4 | 9
Type of surgery [Count of Participants; unit: Participants]
  Knee | 168 | 170 | 338
  Hip | 73 | 75 | 148
Pre-operative opioid [Count of Participants; unit: Participants] | 50 | 57 | 107
Pre-operative Celecoxib [Count of Participants; unit: Participants] | 198 | 195 | 393
Pre-operative Pregabalin [Count of Participants; unit: Participants] | 230 | 232 | 462
Intra-operative total opioid [Median (Inter-Quartile Range); unit: morphine milligram equivalents (MME)] | 10.0 [6.7 to 16.7] | 10.0 [6.7 to 15.0] | 10.0 [6.7 to 15.0]
Intra-operative Ketorolac [Count of Participants; unit: Participants] | 35 | 36 | 71
Intra-operative Bupivacaine Liposome Injectable Suspension [Count of Participants; unit: Participants] | 163 | 162 | 325

OUTCOME MEASURES:

1. Primary Outcome: Total Post-operative Use of Opioids
Description: Post-operative use of opioids, measured in morphine milligram equivalent (MME) units
Time Frame: During post-op period up to 24 hrs after surgery
Measure: Median (Inter-Quartile Range); unit: Morphine milligram equivalents (MME)
Arm/Group | Oral Acetaminophen | IV Acetaminophen
Number analyzed (Participants) | 241 | 245
Morphine milligram equivalents (MME) | 21.7 [12.5 to 33.6] | 21.7 [11.3 to 34.4]

2. Secondary Outcome: Patient-rated Pain in the Post-operative Period
Description: Patient-rated pain in the post-operative period was collected using a 10-point visual analog scale (VAS). A score of 0 indicates no pain; higher scores indicate greater pain. Minimum score for each VAS measurement is 0; Maximum score for each VAS measurement is 10. VAS scores were averaged for each patient.
Time Frame: Standard-of-care post-op assessment intervals during post-op period up to 24 hrs after surgery
Measure: Median (Inter-Quartile Range); unit: Visual analog pain scale (0-10)
Arm/Group | Oral Acetaminophen | IV Acetaminophen
Number analyzed (Participants) | 241 | 245
Visual analog pain scale (0-10) | 3.6 [2.4 to 5.0] | 3.4 [2.1 to 4.8]

3. Other Pre Specified Outcome: Post-operative Nausea and Vomiting
Time Frame: During post-op period up to 24 hrs after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Acetaminophen | IV Acetaminophen
Number analyzed (Participants) | 241 | 245
Participants
  Nausea | 51 | 53
  Vomiting | 19 | 17

4. Other Pre Specified Outcome: Time to First Ambulation - 10 Feet
Time Frame: During post-op period up to 24 hours after surgery
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Oral Acetaminophen | IV Acetaminophen
Number analyzed (Participants) | 241 | 245
Hours | 18.5 [13.8 to 21.3] | 18.8 [15.1 to 21.0]

5. Other Pre Specified Outcome: Time to First Rescue Opioid (PRN Order)
Time Frame: During post-op period up to 24 hrs after surgery
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | Oral Acetaminophen | IV Acetaminophen
Number analyzed (Participants) | 241 | 245
Minutes | 38.0 [20.5 to 151.0] | 41.0 [19.0 to 151.0]

6. Post Hoc Outcome: Post-Anesthesia Care Unit (PACU) Length of Stay, Hours
Description: PACU length of stay was calculated as (PACU discharge moment - PACU admit moment). PACU length of stay is reported in hours.
Time Frame: PACU admission time until PACU discharge time
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Oral Acetaminophen | IV Acetaminophen
Number analyzed (Participants) | 241 | 245
Hours | 2.2 [1.7 to 2.7] | 2.1 [1.7 to 2.6]

7. Post Hoc Outcome: Hospital Length of Stay (LOS)
Description: Total hospital length of stay was calculated as (hospital discharge moment - hospital admission moment). Hospital length of stay is reported in hours.
Time Frame: Pre-op admission to hospital discharge
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Oral Acetaminophen | IV Acetaminophen
Number analyzed (Participants) | 241 | 245
Hours | 58.0 [55.6 to 79.6] | 58.5 [55.5 to 80.9]

ADVERSE EVENTS:
Time Frame: AE/SAE monitoring started at first study drug dose and ended when subjects were discharged from the Post-Anesthesia Care Unit. The time period varied among subjects but was never more than 24 hours total.
Description: Since both the PO and IV forms of the study drug are FDA approved, both are being used within approved labeling, and the study is not being conducted under an Investigational New Drug (IND) application, only events that meet Kettering Health Network's criteria for reporting within the institution's S.A.F.E. reporting system will be reported as SAEs or UPs.
Arm/Group | Oral Acetaminophen | IV Acetaminophen
All-Cause Mortality (participants affected / at risk) | 0/241 | 0/245
Serious Adverse Events (participants affected / at risk) | 0/241 | 0/245
Other Adverse Events (participants affected / at risk) | 0/241 | 0/245

LIMITATIONS AND CAVEATS:
Single hospital, limited to two types of surgical patient. No standard protocol for assessing pain. Oral acetaminophen administered earlier than IV per hospital protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes